CLINICAL TRIAL: NCT03630562
Title: Assay of Pro-angiogenic Cytokines in Exudative Age-Related Macular Degeneration
Acronym: TARMAC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-PP-18
Record Dates: First submitted 2018-01-12; First posted 2018-08-15 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with exudative AMD (Other)
  Interventions: Procedure: Aqueous humor samples collection

INTERVENTIONS:
Procedure: Aqueous humor samples collection — In addition to the routine examinations performed as part of the usual care of AMD patients, an anterior chamber puncture will be performed to collect the aqueous humor samples.

SUMMARY:
Anti-VEGF intravitreal injections are the treatment of choice in age-related macular degeneration (AMD). However 37% of patients are unresponsive or poorly responsive to these therapies. It is still not possible to foresee the patient's response to anti-VEGF injections. A poor response may be related to an activation of alternative pro-angiogenic pathways with over expression of many other pro-angiogenic cytokines.

The primary goal of this study is to measure the aqueous humor concentration of pro-angiogenic cytokines in AMD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of exudative age-related macular degeneration requiring intravitreal anti-VEGF treatment.
* Patient for whom the last intravitreal injection of anti-VEGF in the eye is strictly more than 3 months
* Signature of informed consent
* Affiliation to the French social security system

Exclusion Criteria:

* Pregnant or nursing patient (a urinary pregnancy test will be performed)
* Systemic treatment with anti-VEGF
* Intravitreal treatment with anti-VEGF for less than 3 months regardless of the treated eye.
* Retinal pathology that can modify the secretion of pro-inflammatory cytokines such as diabetic retinopathy, venous occlusions, intermediate and posterior uveitis.
* Diabetes Mellitus
* High Myopia
* Simultaneous participation in another clinical research protocol in exudative AMD
* Person under guardianship, under curatorship, deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Change of pro-angiogenic cytokines concentration in the aqueous humor of patients with exudative AMD at 3 months | At Month 3

SECONDARY OUTCOMES:
Dose of VEGF in the aqueous humor of patients with exudative AMD | At Day 0, Month 1, Month 2, Month 3
Dose of pro inflammatory cytokines in the aqueous humor of patients with exudative AMD | At Day 0, Month 1, Month 2, Month 3
Measurement of visual acuity with Snellen chart | At Day 0, Month 1, Month 2, Month 3
Measurement of visual acuity with ETDRS visual acuity chart | At Day 0, Month 1, Month 2, Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Stéphanie BAILLIF, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital Pasteur 2 - Service d'Ophtalmologie, Nice, France